CLINICAL TRIAL: NCT05692713
Title: Polyomic Biomarker Verification in Adult Chronic Graft-Versus-Host Disease. Applied Biomarkers in Late Effects (ABLE) (ABLE3.0/CTTC2201)
Brief Title: Polyomic Biomarker Verification in Adult Chronic Graft-Versus-Host Disease (ABLE3.0/CTTC2201)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kirk Schultz, Principal Investigator, University of British Columbia
Other Study IDs: H22-03310
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Chronic Graft-versus-Host-Disease; Allogeneic Hematopoietic Stem Cell Transplantation; Leukemia; Blood Cancer; Non-Malignant Hematologic and Lymphocytic Disorder
Keywords: cGvHD; Biomarkers; Blood; Immune cells; Prognostic / diagnostic algorithm; Adult HSC transplant recipients; Blood cancers; Allogeneic HSCT
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Leukemia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood, serum, plasma, cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic graft-versus-host disease (cGvHD) is one of the most serious complications following BMT (Bone Marrow Transplantation). cGvHD occurs when donor immune cells "attack" the tissues and organs of the person receiving the BMT. cGvHD can be difficult to treat once it is established leading to poor quality of life for recipients of a BMT. The goal of this study is to determine if, by using biomarkers, the investigators can predict which patients are at the highest risk of developing cGvHD after BMT, before cGvHD develops.

The ABLE3.0 / CTTC 2201 study will validate and potentially refine the initial predictive biomarker algorithm developed from the original ABLE/PBTMC 1202 study (ABLE1.0), allowing clinicians the ability to pre-emptively predict their patient's future risk of developing both late-acute and chronic GvHD.

This will provide the foundation for the later development of clinical trials aimed at reducing immune suppression quicker after transplant for low-risk patients (<10% risk) and justifying more intensive approaches such as pre-emptive treatments before the onset of chronic GvHD in high-risk patients (>45% risk).

DETAILED DESCRIPTION:
320 adult transplant recipients will be enrolled in this study. The investigators will not recruit healthy participants. Only those undergoing treatments from blood cancers and will be having the transplant procedure will be offered to participate in this study. The control participant group will be determined 12 months post-transplant. This group will consist of those participants who did not develop either chronic or late acute GvHD one year after transplantation.

The investigators will be enrolling allogeneic HCT patients before transplant up through Day -1, following these patients prospectively until 12-months post-transplant for the development of all forms of GvHD - classical acute (aGvHD), late acute (L-aGvHD), and chronic (cGvHD), collecting blood samples and clinical data at day +60, day +100, and at the onset of either L-aGvHD or chronic GvHD (but not classical acute GvHD before day +100). Two more blood samples and clinical data will be collected from transplant recipients who never developed any chronic or late-acute GVHD at the 6- and 12-month post-transplant time points. Case Report Forms (CRFs) will be completed on the REDCap platform.

If chronic GvHD develops at any time after transplant (Day 0 to 1 year), or if any form of GvHD occurs at or after day +100 (whether late acute, chronic GvHD, or overlap syndrome), a blood sample will be drawn before escalating immune suppression, and the onset GvHD case report form will be completed following the protocol. If chronic GvHD is confirmed, an additional CRF will be submitted at 12-months post-transplant to document new cGvHD manifestations, severity, and response to therapy.

A blood sample will not be collected and a CRF will not be completed if classical acute GvHD occurs before Day 100. Staging and grading of classical acute GvHD however will occur on the main case report forms.

On average, patients will have up to 4 blood samples drawn over the course of 1-year post-transplant, depending upon their overall scenario, event and GvHD status.

For clinicians and site PIs, the primary responsibility will be monitoring patients for the development of all forms of GvHD (classical acute, late acute, and chronic GvHD), including accurate documentation, and near real-time reporting of detailed clinical data capture of staging / grading / clinical features /severity and responses to therapy for patients with late-acute and chronic GvHD.

Blood samples drawn from patients will be shipped to the Schultz Laboratory in Vancouver, BC, Canada, processed and analyzed for cGvHD biomarkers. Cell phenotyping by flow cytometry will be carried out on whole blood. Plasma will be used in ELISA, metabolomic analysis and enzymatic assays. Blood cells will be used for B- and T- cell receptors research. A statistical validation of the previously developed pediatric risk predictor in adult population will be be performed based on the estimated overall frequency of cGvHD at 20% or patients.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Any indication for allogeneic hematopoietic stem cell transplant (malignant and nonmalignant);
2. Age >18 years (those who reached the age of majority) at the time of transplant (on Day 0);
3. Any conditioning regimen (including myeloablative or reduced-toxicity/reduced-intensity);
4. Any graft source (bone marrow, peripheral blood, cord blood);
5. Any GvHD prophylaxis strategy, including serotherapy such as ATG or alemtuzumab;
6. Haploidentical transplants, including post-transplant cyclophosphamide and alpha-beta TCR depletion, are allowed

EXCLUSION CRITERIA:

1. Age < 18 years (or under the age of majority) at the time of consent;
2. Second or greater allogeneic transplant;
3. Pure CD34+ selected stem cell grafts (not including C34+ cell enrichment used in alpha-beta TCR depleted haploidentical grafts, which are allowed);
4. Inability of a center to follow a patient for the development of late-acute and chronic GvHD until 1-year post-transplant (referral sites who transplant patients from outside institutions should not enroll participants if sending back to the referring site early, such that long-term follow up, blood, and data collection cannot be assured).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allogeneic Stem Cell Transplant recipients
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Onset of Early cGvHD | Before Day 100 post-transplant
  Early chronic GvHD including overlap syndrome
Onset of cGvHD or L-aGvHD | After Day 100 post-transplant
  Chronic GvHD after Day 100, Late acute GvHD (de-novo or recurrent) after Day 100, or cases of overlap syndrome after Day 100
No cGvHD or L-aGvHD | 12 months post-transplant
  No Chronic or Late-acute GvHD ever develops at any time point in first year post-transplant (regardless of whether or not classical acute GvHD develops in the first 100 days after transplant)

SECONDARY OUTCOMES:
Early Event (criterium for coming off-study) | Before Day 100 post-transplant
  A patient will be taken off study if relapse, mortality, non-engraftment or second transplant occurred

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R. Schultz, MD, Principal Investigator — University of British Columbia / BC Children's Hospital
Locations (10):
- United States (3):
  - Washington University St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oregon Health & Science University, Portland, Oregon
- Canada (7):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - NS Health, Halifax, Nova Scotia
  - Juravinski Hospital & Cancer Centre, Hamilton, Ontario
  - LHSC: Victoria Hospital, London, Ontario
  - UHN Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Québec - Université Laval, Laval, Quebec
  - McGill University Health Center, Montreal, Quebec